CLINICAL TRIAL: NCT06842524
Title: Dihydroartemisinin for the Treatment of Polycystic Ovary Syndrome: a Multi-centre Placebo-controlled Randomized Clinical Trial
Brief Title: Dihydroartemisinin for the Treatment of Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2024-417(2)
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; Dihydroartemisinin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — artenimol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dihydroartemisinin Arm (Active Comparator): Dihydroartemisinin tablets 40mg tid for 90 days
  Interventions: Drug: Dihydroartemisinin
- Placebo Arm (Placebo Comparator): Idential placebo tid for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dihydroartemisinin — Dihydroartemisinin tablets 40mg tid po for 90 days
  Arms: Dihydroartemisinin Arm
Drug: Placebo — Identical placebo tid for 90 days
  Arms: Placebo Arm

SUMMARY:
Polycystic ovarian syndrome (PCOS) is the most frequent endocrine disorder affecting women of reproductive age, with a prevalence of 10 to 13%. PCOS is characterized by irregular menstrual cylcles/ovulatory dysfunction, hyperandrogenism, and polycystic ovarian morphology. For infertile patients seeking ovulation induction, letrozole is the drug of first choice. For PCOS patients not seeking pregnancy, there exists a variety of treatments to alleviate symptoms. It has been demonstrated that artemisinin derivatives can promote energy expenditures and insulin sensitivity by activating thermogenic adipocytes, thereby protecting against diet-induced obesity and metabolic disorders in rodents. Recently, we showed in a single arm pilot study including 19 PCOS-patients, that dihydroartemisinin ameliorated hyperandrogenemia reduced antral follicle count and normalized menstrual cycles. Based on these findings, we aim to evaluate the efficacy of dihydroartemisinin in women with PCOS in a placebo controlled randomized clinical trial. The primary outcome is return of regular menstrual cycles within 6 months after start of treatment, with antral follicle count and metabolic profile being secondary outcomes. The results will potentially impact the standard of care for patients diagnosed with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS defined as having irregular menstrual cycles and hyperandrogenism. Irregular menstrual cycles are defined as < 21 or > 35 days or < 8 cycles per year. Hyperandrogenism refers to either hyperandrogenemia or hirsutism. Hyperandrogenemia will be defined as an elevated total testosterone >1.67 nmol/L measured by Elecsys Testosterone II (Roche Diagnostics). Hirsutism is determined by a modified Ferriman-Gallwey Score >4 at screening exam.
* Body Mass Index (BMI) between 18.5 and 28 kg/M2
* Negative pregnancy test
* No plan for pregnancy in the coming 6 months

Exclusion Criteria:

* Patients on oral contraceptives. A two-month washout period will be required prior to screening for patients on these agents. A one-month washout will be required for patients on oral cyclic progestins. Patients on depo-progestins or hormonal implants are excluded.
* Patients with liver disease defined as ALT or AST above normal range of each participating center, or total bilirubin>30umol/L. Metabolic dysfunction-associated steatotic liver disease (MASLD) with normal ALT and AST can be included.
* Patients with anemia (Hemoglobin < 12 g/dL) or neutropenia (neutrocyte <1.8×10^9/L).
* Patients with renal disease defined as serum creatinine> 115umol/L.
* Patients diagnosed with other endocrine diseases that are known to cause secondary polycystic ovary morphology, e.g., Cushing's syndrome, hyperprolactinemia, congenital adrenal hyperplasia (21-hydroxylase deficiency or other enzyme deficiency), hypothyroidism, etc.
* Patients diagnosed with Type 1 or Type 2 diabetes.
* Patients with known heart disease, like heart failure, atrial fibrillation, coronary heart disease, etc.
* Patients with a history of any type of cancer.
* Patients taking other medications known to affect reproductive function or metabolism. These medications include GnRH agonists and antagonists, antiandrogens, gonadotropins, GLP-1 receptor agonist, SGLT2i, metformin and thiazolidinediones. The washout period on all these medications will be two months.
* Patients who have undergone a bariatric surgery procedure within the past 12 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of a regular menstrual cycle | From the start of treatment to the end of follow-up at 26 weeks
  The occurrence of a regular menstrual cycle is defined as at least three consecutive spontaneous vaginal bleedings lasting for 2-7 days, with intervals between the start of each cycle of 21 and 35 days (inclusive), during the 26-week period after initiating treatment.

SECONDARY OUTCOMES:
The presence of a dominant follicle | From the start of treatment to the end of follow-up at 26 weeks
  This will be verified by transvaginal/transanal ultrasound before predicted ovulation, or testing serum progesterone in the predicted mid-luteal phase (A progesterone level>16nmol/L or 5ng/ml is suggestive of ovulation) in those with at least two consecutive spontaneous bleedings.
The number of bilateral antral follicles | Before and immediately after 90-day treatment
  This will be measured by transvaginal/transanal ultrasound before and immediately after 90-day treatment. Antral follicles are defined as follicles measuring 2-9 mm in diameter in the ovary.
Serum AMH | Before and immediately after 90-day treatment
  This will be measured before and immediately after 90-day treatment.
Serum total testosterone | Before and immediately after 90-day treatment
  This will be measured before and immediately after 90-day treatment.
Serum sex hormone binding globulin (SHBG) | Before and immediately after 90-day treatment
  This will be measured before and immediately after 90-day treatment.
free androgen index (FAI) | Before and immediately after 90-day treatment
  This will be calculated before and immediately after 90-day treatment. FAI is calculated from measurable values for total testosterone and SHBG, using the following equation: FAI = (Total testosterone in nmol/L / SHBG in nmol/L) × 100.
HOMA-IR | Before and immediately after 90-day treatment
  HOMA-IR will be calculated before and immediately after 90-day treatment. HOMA-IR is calculated using the following equation: HOMA-IR = fasting plasma glucose in mmol/L×fasting insulin in μU/ml/22.5.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Dong, MD, Study Chair — Reproductive Medicine Center, Zhongshan Hospital, Fudan University; Xiaoying Li, MD, PhD, Study Director — Department of Endocrinology and Metabolism, Zhongshan Hospital, Fudan University; Jingjing Jiang, MD, PhD, Principal Investigator — Department of Endocrinology and Metabolism, Zhongshan Hospital, Fudan University; Ben Willem Mol, MD, PhD, Principal Investigator — Department of Obstetrics and Gynaecology, Monash University; Wentao Li, MD, PhD, Principal Investigator — National Perinatal Epidemiology and Statistics Unit, Centre for Big Data Research in Health, University of New South Wales
Locations (4):
- China (4):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Women and Children's Hospital, School of Medicine, Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication.
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).